CLINICAL TRIAL: NCT02757365
Title: Efficiency Study of Aspirin to Prevent the Occurrence of Prostate Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yang Lu, Medical Doctor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Huaxi
Record Dates: First submitted 2016-04-18; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: aspirin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aspirin; Levofloxacin

ARMS (4):
- the NSAIDs group (Experimental): Patients in the this Group will received the aspirin 100mg qd until the experiment finished
  Interventions: Drug: aspirin
- the antibiotics group (Experimental): Patients in the this Group will received the Levofloxacin 0.5g qd for 4~8 weeks
  Interventions: Drug: Levofloxacin
- the NSAIDs+antibiotics group (Experimental): Patients in the this Group will received the Levofloxacin 0.5g qd for 4~8 weeks and aspirin 100mg qd until the experiment finished
  Interventions: Drug: aspirin; Drug: Levofloxacin
- the control group (No Intervention): No treatment

INTERVENTIONS:
Drug: aspirin
  Arms: the NSAIDs group; the NSAIDs+antibiotics group
Drug: Levofloxacin
  Arms: the NSAIDs+antibiotics group; the antibiotics group

SUMMARY:
Though the pathogenesis of prostate cancer (PCa) is still obscure, it has been reported, by investigators previous studies and some other researches, that PCa is often combined with tissue inflammation which is closely related to prostate specific antigen (PSA) level. Inflammation could play an important role in the process of occurrence and development of PCa, however the mechanism is unknown. Inflammatory cytokines could not only mediate inflammatory reactions, but also participate in the growth, proliferation, invasion and progression of tumor cells. It has been found that non-steroid anti-inflammatory drugs (NSAIDs), such as aspirin, can effectively prevent several inflammation related tumor, and coincidentally, PCa is also closely associated with inflammation. Moreover, latest researches demonstrated that hormone therapy could induce tissue inflammation in PCa, in which a large quantity of immune B cells were attracted into the focal and then a lot of cytokines, such as IKK-β, NF-κB, were released. These cytokines could inhibit apoptosis and promote the growth of tumor cells, which might be a possible mechanism for long-term inflammatory infiltration inducing the occurrence of PCa and the transformation to castration-resistant prostate cancer (CRPC). Based on these proofs, investigators presume it could be possibly an effective way to prevent the occurrence of PCa and the transformation from androgen-dependent prostate cancer to CRPC by means of long-term oral aspirin. In this study, investigators intend to explore the possible effect of anti-inflammatory therapy on the progress of transformations from inflammation to PCa and from androgen-dependent prostate cancer to CRPC. Investigators plan to conduct both clinical trials in four groups, including the control group, the NSAIDs group, the antibiotics group and the NSAIDs+antibiotics group, and a basic experiment in vitro to assess the effectiveness of anti-inflammatory drugs and elucidate the specific molecular mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Specific Antigen(PSA)>10ng/ml
* Suspected of Prostate Cancer
* Prostate Biopsy showed Benign Prostate Hyperplasia with infiltrated with lymphocytes

Exclusion Criteria:

* Serious Complication:heart disease;respiratory disease;blood disease;
* refused to join the trial
* Disease of hemorrhagic tendency

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
prostate specific antigen（PSA,obtain from blood） | 3 months
  Investigators use this index to screen the patient of prostate cancer.PSA is a reliable index to predict the occurrence of prostate cancer,if PSA>10ng/ml,there is much evidence to suspect prostate cancer
digital rectal examination | 3 months
  Estimation of anal sphincter tone(mild;middle;tight,all the evaluation are reported by the same doctor by inserting index finger into anas to detect the sphincter tone)；prostate's the texture(hard;soft);weather there exist nodule on the prostate,diagnosed by touching the surface of the prostate)
ultrasound of the prostate | 3 month
  the size of prostate(size=0.52* anteroposterior diameter*Left and right diameter*vertical diameter);the change of the findings(compared to the last ultrasound findings);calcification(dense echo)
biopsy of the prostate | 3 month
  confirm the diagnosis;the type of prostate cancer;the classification of inflammation
fPSA | 3 months
  a small part of total PSA;obtain from blood;Investigators use this index to screen the patient of prostate cancer.PSA is a reliable index to predict the occurrence of prostate cancer,if PSA>10ng/ml,there is much evidence to suspect prostate cancer;If fPSA/PSA less than 10%,it is highly suspected being prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- West Hospital of China, Chengdu, Sichuan, China